CLINICAL TRIAL: NCT01685996
Title: Zonisamide Augmentation of Varenicline Treatment for Smoking Cessation
Acronym: 1207
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00074143; R21DA034164 (NIH)
Record Dates: First submitted 2012-09-12; First posted 2012-09-17 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Nicotine Dependence
Keywords: tobacco; smoking cessation; nicotine; cigarettes; nicotine withdrawal
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zonisamide (Experimental): participants will receive zonisamide capsules (up to 300 mg) to take once a day.
  Interventions: Drug: zonisamide
- Placebo (Placebo Comparator): Participants will receive placebo capsules to take once a day
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: zonisamide — In addition to zonisamide vs placebo treatment, varenicline tablets will be dispensed with specific instructions to take at the recommended doses for smoking cessation Participants will receive brief smoking cessation counseling and referral to a quitline
  Other Names: zonegran®
  Arms: zonisamide
Drug: placebo
  Arms: Placebo

SUMMARY:
Randomized trial to evaluate whether zonisamide can enhance varenicline-induced smoking cessation.

DETAILED DESCRIPTION:
About 20.6 % of the US population smokes cigarettes. This group includes nicotine dependent smokers who are resistant to current smoking cessation treatments. Varenicline is a smoking cessation medication found in meta-analytic reviews to be superior to other smoking cessation treatments, but 56% of patients who take varenicline do not quit. One strategy to increase quit rates may be to administer a second medication to augment the efficacy of varenicline. The anti-epileptic medication zonisamide is a good candidate for adjunct treatment as it increases dopaminergic tone, normalizes glutamate homeostasis, potentiates Gamma-Aminobutyric Acid (GABA) release. Zonisamide improves sleep and promotes weight loss, two prominent issues not addressed by varenicline. Finally, the PI of this proposal has documented unpleasant changes in the taste of cigarettes and reductions in nicotine withdrawal among smokers receiving zonisamide as part of another clinical trial. The proposed study will explore the efficacy of varenicline + zonisamide for smoking cessation in a controlled, clinical trial. Eligible participants (n=60) will be smokers (>10 cig/day for >1 year) seeking treatment. They will be randomly assigned to receive varenicline + double-blind zonisamide or placebo for a 10-weeks. Participants will visit the clinic weekly to receive medications and smoking cessation counseling and to complete self-report questionnaires. Smoking status will be assessed via weekly urinalysis testing for cotinine (abstinence: <200ng/ml). Cotinine is a sensitive indicator of smoking status with a longer half-life then carbon monoxide (CO) and is more likely to detect low or intermittent smoking. The study hypothesis is that participants who receive the combination zonisamide + varenicline will achieve greater smoking abstinence compared to varenicline alone. The primary outcome measure will be the 4-week rate of biochemically-confirmed continuous smoking abstinence during weeks 7-10. Secondary outcomes will include self-reported rates of smoking, subjective effects of cigarettes, weight change from baseline to week 10, sleep quality, and nicotine withdrawal severity. This study will advance the science and clinical treatment of smoking cessation, and will provide the prerequisite data to develop a larger scale clinical trial evaluation of the combination zonisamide + varenicline for smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 - 65 years old; smoking > 10 cigarettes per day for > 1 year
* Desire to quit smoking
* Provide a cotinine positive urine sample
* Commitment to come to the clinic once a week for the 10-week study duration

Exclusion Criteria:

* Allergy to varenicline or sulfonamide drugs (e.g., trimethoprim/sulfamethoxazole, zonisamide or topiramate);
* Renal insufficiency (eGFR < 60 mL)
* Renal tubular acidosis
* History of nephrolithiasis
* Unexplained hematuria
* Transaminase elevations > 3 times the Upper Limit of Normal (ULN)
* BMI < 19
* Diabetes mellitus
* Respiratory insufficiency
* Asthma requiring medication
* Heart failure
* Chronic diarrhea predisposing to acidosis
* Glaucoma, family history of glaucoma, one-sided blindness
* History of seizures or use of anticonvulsant medications (not including sedatives)
* HIV infection on HAART medication (or CD4 T cell count < 200 /mL)
* History of serious psychiatric disorder: psychosis, dementia, depression requiring medication in last 6 months, suicidal or homicidal ideation, evidence of violent behavior in the last 6 months.
* Recent use (last 30 days) of bupropion, nortriptyline, or clonidine
* Recent use (last 30 days) of Nicotine Replacement Products that would interfere with urine cotinine testing
* Use of tobacco products other than cigarettes
* For female participants, pregnancy, lactation, or refusal to use an effective method of contraception.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Umbricht, M.D., Principal Investigator — Assistant Professor Behavioral Pharmacology Research Unit The Johns Hopkins University School of Medicine 5510 Nathan Shock Drive Baltimore, MD 21224 tel: 410-550-1917 fax:410-550-0011 annieumbricht@jhu.edu
Locations (1):
- Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Dunn KE, Marcus TF, Kim C, Schroeder JR, Vandrey R, Umbricht A. Zonisamide Reduces Withdrawal Symptoms But Does Not Enhance Varenicline-Induced Smoking Cessation. Nicotine Tob Res. 2016 May;18(5):1171-9. doi: 10.1093/ntr/ntv236. Epub 2015 Oct 17. PMID 26476459

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants will receive placebo capsules to take once a day
  placebo
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 34 | 40
Completed | 18 | 27
Not Completed | 16 | 13

BASELINE CHARACTERISTICS:
Groups:
- Zonisamide: Participants receive zonisamide + varenicline for smoking cessation
- Placebo: Participants receive placebo + varenicline for smoking cessation
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 34 | 40 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (9.8) | 45.9 (9.7) | 45.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 26 | 27 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 34 | 39 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 27 | 50
  White | 11 | 13 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 34 | 40 | 74

OUTCOME MEASURES:

1. Primary Outcome: Percent Participants Abstinent From Smoking During Study Weeks 7-10
Description: Biochemically-verified continuous smoking abstinence during weeks 7-10 of the study.
Time Frame: weeks 7-10
Measure: Count of Participants; unit: Participants
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 34 | 40
Participants | 5 | 6

2. Secondary Outcome: Nicotine Withdrawal Symptom Severity
Description: Total Score from the Minnesota Nicotine Withdrawal Questionnaire (MNWQ), assessed at weekly visits. The MNWQ is a commonly-used 12-item Likert scale self-report measure of nicotine symptoms. Individual symptoms were rated from 0 (none) to 4 (severe) for each item and the Total score range was 0 - 48. Ratings were collected once weekly during study visits.
Time Frame: Past 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 34 | 40
units on a scale
  Screening Visit | 4.6 (6.0) | 5.6 (5.5)
  Admission Visit | 5.1 (5.3) | 7.0 (6.3)
  Week 1 (pre-quit day) | 5.3 (6.) | 6.2 (7.3)
  Week 2 (pre-quit day) | 4.8 (6.0) | 5.7 (6.3)
  Week 3 (target quit day) | 4.7 (5.4) | 6.6 (7.0)
  Week 4 | 3.8 (5.1) | 5.9 (7.0)
  Week 5 | 3.8 (3.7) | 4.7 (5.3)
  Week 6 | 3.4 (4.3) | 4.0 (5.0)
  Week 7 | 3.8 (4.7) | 4.4 (4.7)
  Week 8 | 2.7 (3.3) | 4.0 (4.5)
  Week 9 | 3.1 (3.0) | 4.1 (4.4)
  Week 10 | 2.6 (4.9) | 4.8 (5.8)

ADVERSE EVENTS:
Time Frame: Adverse events were collected systematically during each study visit for the duration of the 10-week study. All events that were rated as being possibly, probably, or definitely related to study participation are reported. Events can represent nicotine withdrawal symptoms (e.g. all events were documented and nicotine withdrawal symptoms were not excluded from Adverse Events (AE) reporting).
Arm/Group | Zonisamide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/40
Other Adverse Events (participants affected / at risk) | 28/34 | 28/40
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zonisamide (N=34) | Placebo (N=40)
Chest Pain (Cardiac disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 5 (5) | 4 (6)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritis (itching) (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Sweating Increased (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (6) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (14) | 11 (14)
Sore Throat (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (4) | 2 (2)
Chemistry Abnormal (Hepatobiliary disorders) | 2 (2) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Jaw Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain Lower Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adjustment Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Change in Mental Status (Psychiatric disorders) | 0 (0) | 1 (1)
Difficulty Concentrating (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Nervous system disorders) | 3 (3) | 1 (1)
Anxiety (Nervous system disorders) | 0 (0) | 3 (3)
Depression (Nervous system disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 3 (3) | 2 (2)
Dream Abnormal (Nervous system disorders) | 8 (9) | 7 (7)
Drowsiness (Nervous system disorders) | 6 (6) | 4 (5)
Fatigue (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Nervous system disorders) | 7 (8) | 3 (3)
Irritability (Nervous system disorders) | 6 (6) | 7 (7)
Paranoid (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 1 (1) | 0 (0)
Restlessness (Nervous system disorders) | 1 (1) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hot Flashes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Itching Eyes (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain- Eye (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No